CLINICAL TRIAL: NCT02680093
Title: Birth Rate in Conservative Monitoring of Pregnancy Beyond the Date of Birth.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0602-15
Record Dates: First submitted 2016-01-21; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Pregnancy, Prolonged
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cervical length in pregnant women.: Pregnant Women beyond the date of birth in conservative monitoring and prenatal follow-up. will be followed while coming to routine monitoring.
  physiological parameter of cervical length will be measured as the differential predictor to determine their due date.
  Interventions: Other: Cervical length in pregnant women.

INTERVENTIONS:
Other: Cervical length in pregnant women. — Pregnant Women beyond the date of birth. will be followed while coming to routine monitoring. physiological parameter of cervical length will be measured as the differential predictor to determine their due date. the cervical length will be measured as part of routine gynecologic examination to women who come for routine over due date follow up.
  additional medical data will be collected from the patient medical record.- demographic data, and all the routine prenatal medical care the women will receive up to the delivery.and delivery out comes.

SUMMARY:
Pregnant Women beyond the date of birth. will be followed while coming to routine monitoring. physiological parameter of cervical length will be measured as the differential predictor to determine their due date. the cervical length will be measured as part of routine gynecologic examination to women who come for routine over due date follow up.

additional medical data will be collected from the patient medical record.- demographic data, and all the routine prenatal medical care the women will receive up to the delivery.and delivery outcomes.

DETAILED DESCRIPTION:
The clinical part of the study: the first visit of pregnancy monitoring is carried out at 40 full weeks. First visit to make sure the gestational age to receive full medical anamnesis , perform physical examination and vaginal and NST and BPP. Also, assess the clinical weight and when the need arises assessment of weight sonography. monitoring fetal movements . The women are ordered to return for routine check ups every 3 days. from - 41 full weeks the women should come every two days and 42 weeks should be referred for induction. In practice, the women offered induction at 41 weeks + 3 or 4 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-50 .
2. Individual fetus
3. The dating of gestational age based on first- trimester ultrasonography or by last menstrual
4. Gestational age between 39 weeks and 0 days to 41 weeks and 6 days .
5. The pregnant women is not in pain ( VAS <3 ) while signing on consent to participate.
6. Normal fetal monitoring measures and Sonar
7. Expectant mother is in active labor
8. Consent to participate

Exclusion Criteria:

1. Multi-pass Pregnancy
2. Without accurate dating of gestational age based on first- trimester ultrasonography or by last menstrual
3. Indicators for abnormal fetal monitoring and / or Sonar
4. Active labor
5. pain ( VAS > = 3 )
6. Expectant mother does not agree to participate or delivery if consent was given earlier

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant Women beyond the date of birth in conservative monitoring and prenatal follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Time interval between measurement of cervical length and delivery | 2 weeks.
  According to our local protocol post date surveillance is stated from 40+0 weeks of gestation. Each gravida undergoes vaginal examination using sonographic measurement of cervical length(in mm) using trans-vaginal sonar.

SECONDARY OUTCOMES:
Delivery with in 48 hours | 48 hours
Delivery with in 7 days | 7 days
Necessity of labor induction duo to post date | 2 weeks
  yes or no. documenting what kind of induction performed.

CONTACTS AND LOCATIONS:
Overall Officials: yariv yogev, professor, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No